CLINICAL TRIAL: NCT05873231
Title: Role of the Gut Microbiome in Anti-tumor Therapy Induced Diarrhea
Acronym: TKI
Status: Recruiting | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 35-015 ex 20/21
Record Dates: First submitted 2023-05-15; First posted 2023-05-24 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum, plasma, urine, stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The role of the gut microbiome in the development of side effects of anti cancer treatment will be assessed in this longitudinal cohort study.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is the 5th most common tumor worldwide and the second most frequent cause of cancer-related death globally. HCC represents about 90% of primary liver cancers and constitutes a major global health problem.Therapeutic approaches depend on the stage of the disease. In the last decade systemic therapy approaches complement surgical and locoregional treatment in advanced disease stages.

The current first-line drug class used to treat locally advanced and metastasized HCC are tyrosine kinase inhibitors (TKIs). At the moment the multikinase inhibitors sorafenib, lenvatinib and regorafenib are licensed in Austria for treatment of HCC: TKIs are a class of small molecule drugs that block the intracellular signals which drive proliferation in many malignant cells by specifically inhibiting the kinase function of individual intracellular pathways involved in receptor-mediated growth signaling.Diarrhea is one of the most common side effects of TKIs, that often prevents optimal dosage and thereby limits efficacy of systemic cancer therapy. Mechanisms of TKI induced diarrhea are largely unknown, speculations span from induction of exocrine pancreatic insufficiency leading to vitamin malabsorption and hypophosphatemia to enterocyte malfunction. Recently, accumulating data suggest that the composition of gut microbiome may also affect efficacy and toxicity of cancer therapy. In a small pilot study (n=25) patients who did not develop diarrhea under TKI had a higher abundance of Butyricimonas and a lower abundance of Citrobacter, Peptostreptococcus, and Staphylococcaceae. To the best of our knowledge, microbiome composition in patients with TKI induced diarrhea has not been studied in detail yet. However, this information is of clinical relevance since the manipulation of the gut microbiota through antibiotics, probiotics, prebiotics or fecal transplantation is an interesting strategy to improve efficacy and mitigate toxicity of anticancer drugs such as TKI. Probiotics for example have been shown to be able to prevent and treat diarrhea and may therefore be a valuable option to prevent or treat TKI-induced side effects.

In 2019 around 5000 Austrian citizens were diagnosed with lung cancer. The diagnosis is associated with a very poor prognosis compared to other malignant diseases. However, the introduction of checkpoint inhibitors has led to a revolutionary improvement in prognosis for those that respond.

Immune-Checkpoints are immunologic pathways that are used by tumor cells to evade destruction by immune cells. The most important checkpoints to date are programmed death ligand 1 (PDL-1), cytotoxic T lymphocyte antigen-4 (CTLA-4) and TIGIT. Antagonization of these check points by monoclonal antibodys can largely improve antineoplastic efficacy of immune cells.

These immune checkpoint inhibitors (ICI) are essential part of modern neoadjuvant, adjuvant and palliative oncologic therapy concepts. ICI-treatment may lead to remarkable responses. However, 60 to 80 percent of patients do not respond to therapy.Although Tumor-PDL-1 level has shown some predictive value and is therefore used in clinical praxis it cannot predict response reliably.

Many preclinical and clinical trials showed evidence of relevant impact of the composition of the microbiome of the gut and response to ICI. Therefore, the microbiome of the gut may be promising biomarker and even possible target for intervention to predict and improve ICI response in the future. However, the exact optimal composition of the gut microbiome and the strategies for intervention are still unclear.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Start of a systemic anti-cancer therapy
* Informed consent

Exclusion Criteria:

* • Pre-existing diarrhoea

  * Antibiotic therapy -4 to -1 week before inclusion
  * Probiotic treatment -4 to -1 week before inclusion
  * Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients receiving systemic anti cancer therapy
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-04-28 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
gut microbiome composition | 4-12 weeks
  16s sequencing

SECONDARY OUTCOMES:
stool zonulin | 4-12 weeks
  ELISA
stool calprotectin | 4-12 weeks
  ELISA
serum lipopolysaccharide binding protein | 4-12 weeks
  ELISA
serum soluble cluster of differentiation (CD)14 | 4-12 weeks
  ELISA
Bristol stool scale (BSS) | 4-12 weeks
  questionnaire on stool consistency and frequency, 1-7, 3-4 is normal
gastrointestinal quality of life (GIQLI) | 4-12 weeks
  questionnaire on gastrointestinal quality of life, 0-144, higher scores are better

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine, Medical University of Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: Yes
Sequencing data will be shared in an open repository
Time Frame: upon publication of the results
Access Criteria: open access